CLINICAL TRIAL: NCT05892250
Title: Effects of Dynamic Humeral Centering Exercises on Functionality and Disability in Subacromial Pain Syndrome
Brief Title: Dynamic Humeral Centering Exercises in Subacromial Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Antofagasta (Other)
Responsible Party: Principal Investigator, Juan Guerrero Henriquez, Principal Investigator, Universidad de Antofagasta
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17798315
Record Dates: First submitted 2023-05-18; First posted 2023-06-07 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Shoulder Pain; Shoulder Impingement Syndrome
MeSH Terms: conditions — Shoulder Pain; Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Intervention will consist of a conventional physical therapy treatment program that includes manual therapy techniques and exercise
  Interventions: Behavioral: Conventional physical therapy
- Experimental group (Experimental): Intervention will consist of a conventional physical therapy treatment program that includes manual therapy techniques and exercise plus Dynamic Humeral Centering exercises
  Interventions: Behavioral: Conventional physical therapy + Dynamic Humeral Centering exercises

INTERVENTIONS:
Behavioral: Conventional physical therapy — Manual techniques and therapeutic exercise
  Arms: Control group
Behavioral: Conventional physical therapy + Dynamic Humeral Centering exercises — Manual techniques and therapeutic exercise and active dynamic humeral centering exercises
  Arms: Experimental group

SUMMARY:
Subacromial pain syndrome is one of the most common musculoskeletal health conditions, causing decreased of range of motion, loss of muscle strength and disability in the shoulder region. It has been proposed that dynamic humeral centering exercises could contribute to overcome these disorders, through the modification of the dimensions of the subacromial space, however, there is no consensus on its effectiveness nor direct variables that account for its efficacy. Therefore, the aim of this research is to determine the effects of a dynamic humeral centering exercise program on the functionality and disability of patients with subacromial pain syndrome.The effects of the dynamic humeral head exercises program, as well as the objective description of factors and variables associated with subacromial pain syndrome, will also allow rehabilitation science professionals to aim their interventions according to the knowledge of direct variables, which will allow objective follow-up of interventions on subacromial pain syndrome diagnosed patients.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old and less than 60 years old.
* Pain in the lateral and upper arm region for more than two weeks of evolution.
* At least three positive tests in the following: Neer's impingement sign, Hawkins-Kennedy impingement sign, Pattes' maneuver, Jobe's test or painful arch.

Exclusion Criteria:

* Having any of the following diagnoses: frozen shoulder, shoulder girdle joint instability, cancer, glenohumeral arthrosis, symptomatic acromioclavicular arthritis, glenohumeral arthritis, rheumatoid arthritis, or fibromyalgia.
* Cervical or thoracic pain.
* Fracture or surgery in the shoulder region or in the last 6 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-07-24 (Estimated); Study Completion 2025-12-18 (Estimated)

PRIMARY OUTCOMES:
Subacromial space dimensions | baseline
  Ultrasonography measure of coracohumeral and acromiohumeral distances

SECONDARY OUTCOMES:
Pain intensity | baseline
  Participants' self-reported pain intensity during activities of daily living, night pain, and pain at rest
Range of motion | baseline
  Active and passive range of motion in coronal, sagital and transverse planes
Muscular endurance | baseline
  Time (in seconds) it takes for the participant to become fatigued when performing repetitive movements with the upper extremity in the frontal plane
Muscular endurance | baseline
  Number of repetitions performed by the subject until fatigue occurs when performing repetitive movements with the upper limb in the frontal plane
Shoulder Pain and Disability Index | baseline
  Measures the percentage of disability in a person, with a minimum value of 0 (best) and a maximum of 100 percent.(worse)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Antofagasta, Antofagasta, Chile

IPD SHARING:
Plan to Share IPD: Yes
The information will be provided to other researchers upon request to the principal investigator of the project.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available once there are publications associated with the clinical trial. These data will be available for 4 years.
Access Criteria: By e-mail request